CLINICAL TRIAL: NCT03423576
Title: Effects of a Comprehensive Patient-centered Health Service With a Focus on Psychosocial Services for Patients With Rare Diseases Using Cystic Fibrosis as an Example (Evaluation Eines Ganzheitlichen Patientenzentrierten Versorgungsmodells für Patienten Mit Seltenen Erkrankungen Unter Besonderer Berücksichtigung Der Psychosozialen Versorgung am Beispiel Mukoviszidose)
Brief Title: Effects of a Comprehensive Patient-centered Health Service in Cystic Fibrosis (VEMSE-CF)
Acronym: VEMSE-CF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mukoviszidose Institut gGmbH (Other)
Collaborators: Federal Ministry of Health, Germany (Other Government); Wuerzburg University Hospital (Other); Hannover Medical School (Other); Goethe University (Other); CF-Center Hamburg-Altona (Unknown); University Hospital Ulm (Other); Medical Association of Lower Saxony (Ärztekammer Niedersachsen), Germany (Unknown)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Purpose: Health Services Research
Other Study IDs: VEMSE-CF
Record Dates: First submitted 2018-01-23; First posted 2018-02-06 (Actual); Last update posted 2018-02-19 (Actual); Status verified 2018-02

CONDITIONS: Cystic Fibrosis
Keywords: health services; FEV1; BMI; quality of life; mental stress
MeSH Terms: conditions — Cystic Fibrosis; Stress, Psychological | interventions — Methods

STUDY DESIGN:
Masking Description: there was no masking of patients or outcome assessors
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): comprehensive patient-centered outpatient health service with multiple components. These components included the addition of a case-manager, structured interventions to improve patient education and adherence to therapy, psychological counselling, social services, and exercise advice. For each Patient, relevant components were identified and a written Intervention plan was negotiated and signed.
  Interventions: Behavioral: comprehensive patient-centered outpatient health service with multiple components
- Control (No Intervention): Standard care

INTERVENTIONS:
Behavioral: comprehensive patient-centered outpatient health service with multiple components — Individualized multi-component education and counselling program coordinated by a case Manager.
  Other Names: Intervention
  Arms: Intervention

SUMMARY:
For the Project VEMSE-CF, a comprehensive patient-centered outpatient health service model was developed offering focused interventions in different areas. These included patient education, as well as nutritional and exercise counselling. Special emphasis was given to the psycho-social services. The implementation was supported by a case manager. The model was implemented in three German CF-Centers. For evaluation, Patient data from 13 additional German CF-Centers offering standard care was used as comparison. In total, 153 patients in the Intervention Group and 163 control patients aged 5-52 years contributed data. The primary endpoint was the number of BMI- and FEV1-measurements over 24 months. Secondary endpoints included mortality, lung transplantation, FEV1, BMI, adherence to therapy, Quality of life, and mental stress.

ELIGIBILITY:
Inclusion Criteria:

* confirmed diagnosis of Cystic Fibrosis - written informed consent
* intervention group: care in one of the 3 CF-centers
* control group: care in one of the 13 control CF-centers

Exclusion Criteria:

* post lung Transplantation
* listed for lung Transplantation and planned inpatient stay for more than 4 weeks

Min Age: 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 318 (Actual)
Dates: Start 2011-08-01 (Actual); Primary Completion 2016-02-28 (Actual); Study Completion 2016-12-31 (Actual)

PRIMARY OUTCOMES:
Number of BMI and FEV1 assessments | 24 months
  crude number of assessments (BMI and FEV1) performed during the study period

SECONDARY OUTCOMES:
Mortality | 24 months
  Number of patients deceased during the study period
Referrals for Lung Transplantation | 24 months
  number of patients referred for lung Transplantation during the study
Delta FEV1 | 24 months
  Change in FEV1 from baseline to end of study
Delta BMI | 24 months
  Change in BMI from baseline to end of study
Outpatient visits | 24 months
  Number of outpatient visits during study period
Hospitalizations | 24 months
  number of hospitalizations during the study period

OTHER OUTCOMES:
Delta Proportion of patients with subnormal FEV1 | 24 months
  Change in the Proportion of patients with an FEV1<80% predicted
Delta Proportion of Patients with well preserved BMI | 24 months
  Change in the Proportion of patients with a BMI equal or greater 22 kg/m2 (females) or 23 kg/m2 (males)
Adherence to therapy | 24 months
  Performance of planned assessments (four per year; eight during intervention)
Quality of Life (patients) | 24 months
  Self- or proxy-Report of patients´ Quality of Life: questionnaire - EQ5D (adults) / EQ5D - Y (13-18) / CFQ-R-6-12; three assessments during intervention (begin / after 12 month /after 24 month)
Quality of Life (parents) | 24 months
  self-report of parents´ Quality of Life; questionnaire - EY5D; three assessments during intervention(begin / after 12 month /after 24 month)
Emotional stress (Patients) | 24 months
  Self- or proxy-Report of patients´ emotional stress; questionnaire - Hospital Anxiety and Depression Scale (HADS); three assessments during Intervention (begin / after 12 month /after 24 month)

CONTACTS AND LOCATIONS:
Overall Officials: Uta Düesberg, Dr., Study Chair — Mukoviszidose Institut gGmbH; Miriam Schlangen, Dr., Study Director — Mukoviszidose Institut gGmbH; Lutz Goldbeck, Prof. Dr., Principal Investigator — Ulm University Hospital; Helge Hebestreit, Prof. Dr., Principal Investigator — Wuerzburg University Hospital
Locations (1):
- Mukoviszidose Institut, Bonn, Germany

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Besier T, Born A, Henrich G, Hinz A, Quittner AL, Goldbeck L; TIDES Study Group. Anxiety, depression, and life satisfaction in parents caring for children with cystic fibrosis. Pediatr Pulmonol. 2011 Jul;46(7):672-82. doi: 10.1002/ppul.21423. Epub 2011 Mar 7. PMID 21384564
- [Background] Goldbeck L, Besier T, Hinz A, Singer S, Quittner AL; TIDES Group. Prevalence of symptoms of anxiety and depression in German patients with cystic fibrosis. Chest. 2010 Oct;138(4):929-36. doi: 10.1378/chest.09-2940. Epub 2010 May 14. PMID 20472857
- [Background] Kerem E, Conway S, Elborn S, Heijerman H; Consensus Committee. Standards of care for patients with cystic fibrosis: a European consensus. J Cyst Fibros. 2005 Mar;4(1):7-26. doi: 10.1016/j.jcf.2004.12.002. No abstract available. PMID 15752677
- [Background] Ravens-Sieberer U, Otto C, Kriston L, Rothenberger A, Dopfner M, Herpertz-Dahlmann B, Barkmann C, Schon G, Holling H, Schulte-Markwort M, Klasen F; BELLA study group. The longitudinal BELLA study: design, methods and first results on the course of mental health problems. Eur Child Adolesc Psychiatry. 2015 Jun;24(6):651-63. doi: 10.1007/s00787-014-0638-4. Epub 2014 Nov 27. PMID 25428179
- [Background] Ruf K, Winkler B, Hebestreit A, Gruber W, Hebestreit H. Risks associated with exercise testing and sports participation in cystic fibrosis. J Cyst Fibros. 2010 Sep;9(5):339-45. doi: 10.1016/j.jcf.2010.05.006. Epub 2010 Jul 2. PMID 20584632
- [Background] Sens B, Stern M. (2012) (Hrsg).Qualitätssicherung Mukoviszidose. Überblick über den Gesundheitszustand der Patienten in Deutschland 2012, Bonn/Hannover
- [Background] Graf von der Schulenburg JM, Greiner W, Jost F, Klusen N, Kubin M, Leidl R, Mittendorf T, Rebscher H, Schoeffski O, Vauth C, Volmer T, Wahler S, Wasem J, Weber C; Hanover Consensus Group. German recommendations on health economic evaluation: third and updated version of the Hanover Consensus. Value Health. 2008 Jul-Aug;11(4):539-44. doi: 10.1111/j.1524-4733.2007.00301.x. Epub 2008 Jan 11. No abstract available. PMID 18194408